CLINICAL TRIAL: NCT03931681
Title: A Phase 1 Study of OKI-179 as a Single Agent in Patients With Advanced Solid Tumors
Brief Title: A Study of OKI-179 in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OnKure, Inc. (Industry)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OKI-179-101
Record Dates: First submitted 2019-04-17; First posted 2019-04-30 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: Phase 1 - Dose Escalation (Experimental): Dose escalation trial evaluating OKI-179 given orally on a daily basis. Patients will take OKI-179 orally (PO) on Days 1 - 4, 8 - 11 and 15 - 18 in 21-day cycles (± 3 days), under fasted conditions. The design is a modified 3+3 design to determine the maximum tolerated dose and allows for additional cohorts enrolling subjects with an alternative dosing schedule such as OKI-179 orally (PO) daily on Days 1 - 5, 8 - 12 and 15 - 19 per 21-day cycles or Days 1 - 21 per 21-day cycles to determine the maximum tolerated dose for continuous daily dosing.
  Interventions: Drug: OKI-179

INTERVENTIONS:
Drug: OKI-179 — OKI-179 single agent

SUMMARY:
This study is a Phase 1, single center, open-label study, assessing single agent dose escalation of OKI-179.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria to be eligible for enrollment.

* Histologically or cytologically confirmed solid tumors, advanced or metastatic disease, refractory to standard therapy or for whom no standard therapy exists, or the patient is ineligible for standard therapy(ies).
* At least 1 measurable lesion based on Response Evaluation Criteria in Solid Tumor (RECIST) version 1.1.
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) ≤ 1 within 14 days prior to Cycle 1 Day 1.
* Signed informed consent prior to initiation of any study-related procedures that are not considered standard of care.
* Male or female, ≥ 18 years of age at time of signing consent.
* Adequate hematologic and organ function as defined by the following criteria within 14 days prior to Cycle 1 Day 1:
* Absolute neutrophil count (ANC) ≥ 1.5 × 109/L; excluding measurements obtained within 7 days after daily administration of filgrastim/sargramostim or within 3 weeks after administration of pegfilgrastim.
* Platelet count ≥ 100 × 109/L; excluding measurements obtained within 3 days after transfusion of platelets.
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × upper limits of normal (ULN); if liver function abnormalities are due to underlying liver metastases, AST and ALT ≤ 5 × ULN.
* Total serum bilirubin ≤ 1.5 × ULN, or ≤ 3 × ULN if attributed to Gilbert's Syndrome.
* Serum creatinine ≤ 1.5 x ULN or Creatinine clearance (CrCl) ≥ 50 mL/min; the CrCl can be measured from urine or calculated from serum creatinine (Cockcroft-Gault Equation).
* Female patients of childbearing potential must have a negative serum beta-human chorionic gonadotropin (β-hCG) test within 14 days prior to Cycle 1 Day 1.
* Male patients and female patients of childbearing potential must agree to use an effective method of contraception per institutional standard prior to the first dose and for 90 days after the last dose of OKI-179.
* Willingness and ability to comply with all scheduled visits, treatment plan, laboratory tests and other study procedures.

Exclusion Criteria:

Patients meeting any of the following criteria are ineligible for enrollment in the study:

* Any of the following treatment interventions within the specified time frame prior to Cycle 1 Day 1:
* Major surgery within 28 days (the surgical incision should be fully healed prior to study drug administration).
* Radiation therapy within 21 days; however, if the radiation portal covered ≤ 5% of the bone marrow reserve, the patient is eligible irrespective of the end date of radiotherapy. None of the recently irradiated lesions can be included in the measurable disease assessment.
* Cytotoxic therapy within 21 days (nitrosoureas or mitomycin within 42 days, capecitabine within 14 days).
* Monoclonal antibodies within 28 days.
* Current use of an investigational agent that is not expected to be cleared by Cycle 1 Day 1.

Note: Continuation of luteinizing hormone-releasing hormone (LHRH) agonists for prostate cancer, bisphosphonates or denosumab for bone metastases.

* Side effects from prior treatment interventions not resolved to a Grade ≤ 1 (except alopecia or peripheral neuropathy).
* Prior Histone deacetylase (HDAC), pan-deacetylase (DAC), heat shock protein 90 (HSP90) inhibitors or valproic acid for the treatment of cancer.
* Concomitant malignancies or previous malignancies with less than a 2-year disease free interval at the time of enrollment. Patients with adequately resected basal or squamous cell carcinoma of the skin, carcinoma in situ of the cervix or breast, or Stage 1 prostate cancer or others deemed to be cured by surgery alone or surgery plus radiotherapy in the judgment of the Investigator may enroll irrespective of the time of diagnosis.
* Medical, psychiatric, cognitive, or other conditions that compromise the patient's ability to understand the patient information, to give informed consent, to comply with the study protocol, or to complete the study.
* Any severe concurrent disease or condition (including active systemic infection requiring systemic therapy, uncontrolled diabetes mellitus, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, or cardiac arrhythmia) which, in the judgment of the Investigator, would make the patient inappropriate for study participation.
* Known symptomatic active central nervous system (CNS) metastases and/or carcinomatous meningitis. Stable doses of corticosteroids for at least 2 weeks prior to enrollment for brain metastasis is allowed.
* Significant gastrointestinal abnormalities, including an inability to take oral medication, requirement for IV alimentation, active peptic ulcer, chronic diarrhea or vomiting considered to be clinically significant in the judgment of the Investigator, or prior surgical procedures affecting absorption.
* Known positive serology for the human immunodeficiency virus (HIV) (HIV 1/2 antibodies) or acquired immunodeficiency syndrome (AIDS)-related illness, and/or known active hepatitis B (e.g., hepatitis B surface antigen-reactive) or hepatitis C (e.g., hepatitis C virus ribonucleic acid [qualitative]).
* Pregnant or lactating females.
* 12-lead electrocardiography (ECG) demonstrating a QT interval corrected for heart rate using Fridericia's formula (QTcF) of ≥ 480 msec for males and ≥ 480 msec for females (mean of the triplicate ECG measurements), with the exception for patients with an atrioventricular pacemaker or other conditions (e.g., right bundle branch block) that render the QT measurement invalid.
* History or current evidence of congenital long QT syndrome.
* Taking medications that lead to significant QT prolongation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-05-08 (Actual); Primary Completion 2021-11-27 (Actual); Study Completion 2021-11-27 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) | 2 years
  Tolerability
Determine the safety of the drug according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 5 | 2 years
  * Incidence and severity of adverse events (AEs), graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 5
  * Incidence and severity of Serious Adverse Events
  * Incidence and severity of dose-limiting toxicities (DLTs)
  * Findings of changes in clinical laboratory abnormalities
  * Changes in triplicate 12-lead electrocardiogram (ECG) parameters
  * Changes in the Eastern Cooperative Oncology Group (ECOG) performance status (PS)
  * Changes in physical examination findings

SECONDARY OUTCOMES:
Maximum Concentration (Cmax) of OKI-179 and OKI-006 in Plasma | 2 years
  Plasma concentrations of OKI-179 and OKI-006 will be measured to determine the maximum observed concentration for each compound.
Area Under the Curve (AUC) for OKI-179 and OKI-006 in Plasma | 2 years
  Plasma concentrations of OKI-179 and OKI-006 will be measured to determine the AUC for each compound.
Area Under the Curve (AUC) for OKI-179 and OKI-006 in Urine | 2 years
  Urine concentrations of OKI-179 and OKI-006 will be measured to determine the AUC for each compound.
Time to Maximum Concentration (Tmax) for OKI-179 and OKI-006 in Plasma | 2 years
  Plasma concentrations of OKI-179 and OKI-006 will be measured to determine the Tmax for each compound.
Time to Maximum Concentration (Tmax) for OKI-179 and OKI-006 in Urine | 2 years
  Urine concentrations of OKI-179 and OKI-006 will be measured to determine the Tmax for each compound.
Efficacy as measured by periodic CT/MRI scans using the revised Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1 | 2 years
  * Fraction of patients who have a Complete Response
  * Fraction of patients who have a Partial Response
  * Duration of response (DOR)
  * Progression free survival
  * Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Diamond, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Cancer Center, Aurora, Colorado, United States